CLINICAL TRIAL: NCT04774458
Title: The Safety and Clinical Utilities of the Fluoroscopy-guided Cervical Epidural Approach Using the Contralateral Oblique View: a Prospective Observational Study
Brief Title: Prospective Observation of the Fluoroscopy-guided Cervical Epidural Approach Using the Contralateral Oblique View
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Doo-Hwan Kim, Assistant professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0197
Record Dates: First submitted 2021-02-21; First posted 2021-03-01 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Cervical Intervertebral Disc Disease; Cervical Spinal Stenosis; Cervical Radicular Pain; Herpes Zoster; Postherpetic Neuralgia
Keywords: fluoroscopy; contralateral oblique view; cervical epidural block; cervical epidural space
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluoroscopic-guided cervical epidural access (Experimental): Cervical epidural access with loss of resistance technique using CLO view at 50 degree under fluoroscopic guidance.
  Interventions: Procedure: Fluoroscopic-guided cervical epidural access

INTERVENTIONS:
Procedure: Fluoroscopic-guided cervical epidural access — After identifying the target level of the cervical spine under a fluoroscopy-guided anteroposterior image, an 18-Tuohy needle is inserted through a paramedian approach after local infiltration with 1% lidocaine. When feeling a strong resistance through the needle by a ligamentum flavum, the image intensifier is rotated to 50 degrees contralateral oblique (CLO) direction. After then, the needle is advanced to just before the ventral interlaminar line in CLO view. It is subsequently advanced further until it is in the epidural space using a LOR-to-air technique. Correct epidural access is confirmed by the injection of contrast medium. After identifying epidural space in AP and CLO view without abnormal dispersion of contrast,(vascular uptake, intrathecal spreads, etc.), a 3-4ml mixture of 0.5% lidocaine with dexamethasone 5mg is injected.

SUMMARY:
The aim of the present study is to investigate the safety and clinical utility of contralateral oblique view for fluoroscopic guided cervical epidural access.

DETAILED DESCRIPTION:
A cervical epidural block is a widely used intervention to reduce pain in patients with cervicalgia or cervical radicular pain. To achieve a successful procedure, accurate access to the cervical epidural space is needed. However, careful attention is required for this cervical epidural procedure due to a possibility of serious complications such as spinal cord infarction and quadriplegia due to blood vessel damage, convulsion due to an intravascular drug administration, cerebral infarction due to vascular embolism, subdural or subarachnoid injection, hematoma, and spinal cord injury. Although the use of fluoroscopy improves the safety and accuracy of cervical epidural access, this technique still has significant drawbacks, such as false loss of resistance and difficulty in assessing the depth of the needle tip in lateral views in relation to the epidural space. To overcome this issue, cervical epidural access using the contralateral oblique (CLO) view has been introduced and the ideal angle of CLO view for the cervical spine is reported as 50 degrees.

However, it has not been reported on the safety and clinical utility of using the CLO view during cervical epidural access. Therefore, the investigators planned this study to observe the safety and clinical utility of the CLO view at 50 degrees for the cervical epidural block.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need an epidural space access at C6-7 or C7-T1 level
* Patients who are expected to undergo cervical epidural block
* Patients who are expected to undergo cervical epidural neuroplasty
* 20 ≤ age <80
* When obtaining informed consent voluntarily

Exclusion Criteria:

* Allergy to local anesthetics and contrast dye, and steroid
* Use of anticoagulants or antiplatelet medication, coagulopathy
* Infection at the insertion site
* Neurological or psychiatric disorders
* Prior spine instrumentation
* Pregnancy
* Not visible epidural space due to severe cervical spinal canal stenosis

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Dural puncture event - major complication | Immediately after contrast medium administration during the procedure
  whether a dural puncture event occurs or not during the cervical epidural access

SECONDARY OUTCOMES:
Other complications | Immediately after procedure
  intravascular entry, subdural entry, vasovagal reaction, spinal cord injury
Needling time | Immediately after procedure
  time to access the epidural space after skin insertion
First attempt success | Immediately after procedure
  whether an cervical epidural access is successful at once without any withdrawal of the needle or not
Total number of needle passes | Immediately after procedure
  A needle pass is considered as an advancement of the needle without any withdrawal. If the needle is re-advanced after a withdrawal, it is considered as an additional(second) needle pass.
Rate of success or failure | Immediately after procedure
  Success is defined when contrast medium spreads appropriately in epidural space after physician successfully access cervical epidural space.
Needle tip visualization | One day after the procedure
  The clarity of the needle tip was subjectively graded as 1 (clearly visualized without ambiguity), 2 (poorly visualized or visualized with effort), or 3 (not visualized).
Needle tips location | One day after the procedure
  Location of the needle tip was defined as being significantly before the VILL(Ventral interlaminar line) (-2), just before the VILL (-1), on the VILL (0), just after the VILL (+1), or significantly after the VILL (+2)
False positive/negative loss of resistance | Immediately after procedure
  False positive: Not reaching epidural space despite feeling loss of resistance/ false negative: Reaching epidural space despite not feeling loss of resistance
Post-procedural complication | Up to one month after the procedure
  epidural hematoma, spinal cord injury, infection, abscess, facial flushing, post-dural puncture headache
Radiation dose (cGy) | Immediately after procedure
  Radiation dose (cGy)
Numerical rating scales (NRS) | One month after the procedure
  One month after the procedure, the pain intensity is assessed using a numeric rating scale (0: no pain, 10: unbearable pain).
Global perceived effect (GPE) | One month after the procedure
  One month after the procedure, Patient satisfaction is assessed using global perceived effects on a 7-point scale (GPE). (1: very dissatisfied, 7: very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Hwan Kim, MD, PhD, Principal Investigator — Assistant professor
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Kwon HJ, Kim CS, Kim J, Kim S, Shin JY, Choi SS, Shin JW, Kim DH. Contralateral oblique view can prevent dural puncture in fluoroscopy-guided cervical epidural access: a prospective observational study. Reg Anesth Pain Med. 2023 Dec;48(12):588-593. doi: 10.1136/rapm-2022-104297. Epub 2023 Apr 6. PMID 37024268